CLINICAL TRIAL: NCT00498706
Title: Telephone Versus Face-to-Face Administration of CBT for Depression
Brief Title: Effectiveness of Telephone Versus Face-to-Face CBT in Treating People With Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Mohr, Professor, National Institute of Mental Health (NIMH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH059708 (NIH); R01MH059708 (NIH)
Record Dates: First submitted 2007-07-08; First posted 2007-07-10 (Estimated); Results first posted 2013-07-17 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Depression
Keywords: Depressive Disorder, Major; Cognitive Behavioral Therapy; Psychotherapy; Telemedicine; Primary Care
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telephone-administered CBT (Experimental): Participants will receive telephone-administered cognitive behavioral therapy.
  Interventions: Behavioral: Telephone-administered cognitive behavioral therapy (T-CBT)
- Face-to-face CBT (Active Comparator): Participants will receive face-to-face cognitive behavioral therapy.
  Interventions: Behavioral: Face-to-face administered CBT (FtF-CBT)

INTERVENTIONS:
Behavioral: Telephone-administered cognitive behavioral therapy (T-CBT) — Over 18 weeks, participants will receive eighteen 45-minute sessions of T-CBT administered by a therapist. Participants will undergo telephone-administered sessions twice a week for 2 weeks, once a week for 12 weeks, and once every 2 weeks for the last 4 weeks. Participants will be taught ways to modify thoughts and behaviors that contribute to their depression and ways to maintain the lifestyle changes that they have made.
  Arms: Telephone-administered CBT
Behavioral: Face-to-face administered CBT (FtF-CBT) — Over 18 weeks, participants will receive eighteen 45-minute sessions of FtF-CBT administered by a therapist. Participants will undergo face-to-face administered sessions twice a week for 2 weeks, once a week for 12 weeks, and once every 2 weeks for the last 4 weeks. Participants will be taught ways to modify thoughts and behaviors that contribute to their depression and ways to maintain the lifestyle changes that they have made.
  Arms: Face-to-face CBT

SUMMARY:
This study will compare the effectiveness of telephone versus face-to-face administration of cognitive behavioral therapy in treating people with depression.

DETAILED DESCRIPTION:
Major depressive disorder is a common and often long-lasting disorder with 12-month prevalence rates estimated to be between 6.6% and 10.3%. Although the personal and societal costs of depression are high, it is well established that depression can be effectively treated using antidepressant medication and/or forms of psychotherapy. Several studies have found that when given a choice, about two-thirds of depressed patients prefer psychotherapy or counseling over antidepressant medication. However, a variety of barriers exist to initiating and maintaining psychotherapy. Only about 20% of all patients referred for psychotherapy actually initiate treatment, and of those who do initiate treatment, nearly half drop out before completing treatment. The use of the telephone to deliver treatment services has been recommended as a way to reduce many of the barriers associated with failure to initiate and sustain treatment. When administered over the telephone, cognitive behavioral therapy (CBT), a form of psychotherapy that teaches ways to modify thoughts and behaviors that contribute to depression, may be superior to face-to-face CBT in improving treatment adherence and reducing depressive symptoms. This study will compare the effectiveness of telephone CBT (T-CBT) versus face-to-face CBT (FtF-CBT) in treating people with depression.

Participation in this study will include 18 weeks of treatment and 12 months of follow-up. All participants will first undergo baseline assessments that will include a telephone interview and questionnaires about mood. Participants will then be assigned randomly to receive T-CBT or FtF-CBT. Participants in both groups will receive eighteen 45-minute sessions of their assigned treatment over 18 weeks. Sessions will occur twice a week for 2 weeks, once a week for 12 weeks, and once every 2 weeks for the last 4 weeks. During sessions, participants will learn ways to modify thoughts and behaviors that contribute to their depression and ways to maintain the lifestyle changes that they have made. Treatment sessions will be identical for both groups, except one group will receive sessions over the telephone and the other in-person at a study office. All participants will repeat the baseline assessments at Weeks 4, 9, 14, and 18 of treatment and Months 3, 6, 9, and 12 of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Has a current diagnosis of major depressive disorder
* Has a primary care physician at Northwestern University in Illinois, or one of a number of approved community clinics in Chicago.
* Resides in Illinois
* Has a telephone
* Speaks and reads English

Exclusion Criteria:

* Hearing, voice, or visual impairment
* Meets criteria for dementia
* Diagnosed with a psychotic disorder, bipolar disorder, dissociative disorder, current substance abuse, or other condition for which participation in a clinical trial of psychotherapy may be either inappropriate or dangerous
* Currently receiving individual psychotherapy or planning to receive psychotherapy during the treatment phase of the study
* Planning to be out of town or unavailable for treatment for 4 weeks or more during the scheduled treatment time
* Recent history of suicide attempts or is severely suicidal
* Initiated treatment with an antidepressant in the 2 months before study entry (antidepressant medication is not exclusionary)
* Depression determined to be primarily of an organic etiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2007-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C. Mohr, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Mohr DC, Ho J, Duffecy J, Reifler D, Sokol L, Burns MN, Jin L, Siddique J. Effect of telephone-administered vs face-to-face cognitive behavioral therapy on adherence to therapy and depression outcomes among primary care patients: a randomized trial. JAMA. 2012 Jun 6;307(21):2278-85. doi: 10.1001/jama.2012.5588. PMID 22706833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from November 2007 to December 2010 from general internal medicine clinics in Northwestern Medical Faculty Foundation and Northwestern Memorial Physician's Group, and from 4 primary care clinic members of Northwestern's Practice-Based Research Network.
Period: Overall Study
Arm/Group | Telephone-administered CBT | Face-to-face CBT
Started | 163 | 162
Post Treatment Week 18 | 163 | 162
Completed | 163 | 162
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telephone-administered CBT | Face-to-face CBT | Total
Number analyzed (Participants) | 163 | 162 | 325
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 150 | 148 | 298
  >=65 years | 13 | 14 | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 47.8 (12.6) | 47.5 (13.5) | 47.6 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 127 | 252
  Male | 38 | 35 | 73
Region of Enrollment [Number; unit: participants]
  United States | 163 | 162 | 325

OUTCOME MEASURES:

1. Primary Outcome: Attrition (Number of Therapy Sessions Attended)
Description: Number of therapy sessions attended was collected. At the end of treatment, the total number of sessions attended by each patient was collected.
Time Frame: Post treatment, up to 18 weeks
Population: A randomized controlled trial of 325 Chicago area primary care patients with major depressive disorder, recruited from November 1007 to December 2010.
Measure: Mean (Standard Deviation); unit: Number of Sessions
Units Other Than Participants: sessions
Arm/Group | Telephone-administered CBT | Face-to-face CBT
Number analyzed (Participants) | 163 | 162
Number analyzed (sessions) | 2518 | 2221
Number of Sessions | 15.4 (4.4) | 13.7 (6.1)
Statistical Analysis 1: Comparison: Telephone-administered CBT vs Face-to-face CBT; Test type: Superiority or Other; p = 0.003, t-test, 2 sided; t value = -2.95

2. Primary Outcome: Number of Participants Who Dropped Out of Therapy
Description: Using the number of therapy sessions attended, we categorized patients into:
  1. those who discontinued treatment before session 18, and those who completed session 18.
  2. those who discontinued before Session 5, and those who continued.
Time Frame: Post treatment, up to 18 weeks
Measure: Number; unit: participants
Groups:
- Telephone-administered Cognitive Behavioral Therapy: Participants will receive telephone-administered cognitive behavioral therapy.
- Face-to-face Cognitive Behavioral Therapy: Participants will receive face-to-face cognitive behavioral therapy.
Arm/Group | Telephone-administered Cognitive Behavioral Therapy | Face-to-face Cognitive Behavioral Therapy
Number analyzed (Participants) | 163 | 162
participants
  those who discontinued treatment before session 18 | 34 | 53
  those who discontinued before Session 5, | 7 | 21
Statistical Analysis 1: Comparison: Telephone-administered Cognitive Behavioral Therapy vs Face-to-face Cognitive Behavioral Therapy; Test type: Superiority or Other; p = 0.02, Chi-squared; Chi-square = 5.83
Statistical Analysis 2: Comparison: Telephone-administered Cognitive Behavioral Therapy vs Face-to-face Cognitive Behavioral Therapy; Test type: Superiority or Other; p = .006, Chi-squared; Chi-square = 7.75 — Attrition before week 5 was significantly lower in T-CBT than in face-to-face CBT

3. Secondary Outcome: Health-related Quality of Life (SF-36V), Patient Satisfaction (Satisfaction Index - Mental Health), and Therapeutic Alliance (Working Alliance Inventory - Short Form)
Time Frame: Measured at baseline; Weeks 4, 9, 14, and 18; and Months 3, 6, 9, and 12 of follow-up
Reporting Status: Not Posted

4. Primary Outcome: Patient Health Questionnaire (PHQ)-9
Description: Measures depression on a 9 - item scale. Scores range from 0-27, with 0 being no symptoms. A difference of 5 or more points on the PHQ-9 is considered a clinically meaningful response to treatment.
Time Frame: Measured at baseline; Weeks 4, 9, 14, and 18; and Months 3, 6 post-treatment follow-up
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Telephone-administered CBT | Face-to-face CBT
Number analyzed (Participants) | 162 | 163
units on a scale
  Baseline | 16.76 (4.7) [16.24 to 17.29] | 16.76 (4.8) [16.24 to 17.29]
  Week04 | 10.78 [9.92 to 11.64] | 10.09 [9.21 to 10.97]
  Week09 | 9.05 [8.13 to 9.96] | 8.62 [7.64 to 9.59]
  Week14 | 8.55 [7.53 to 9.56] | 7.77 [6.73 to 8.82]
  Week18 | 6.65 [5.72 to 7.58] | 6.74 [5.74 to 7.73]
  3-month follow-up | 7.59 [6.60 to 8.58] | 6.60 [5.56 to 7.64]
  6-month follow-up | 8.42 [7.38 to 9.46] | 6.30 [5.24 to 7.37]
Statistical Analysis 1: Comparison: Telephone-administered CBT vs Face-to-face CBT; Longitudinal depression scores were modeled with repeated-measures linear regression models.Time was treated as a categorical variable to account for nonlinear effects of time, and an unstructured covariance matrix was assumed; Test type: Non-Inferiority or Equivalence — Noninferiority is established by showing that the true difference between 2 treatment arms is likely to be smaller than a prespecified noninferiority margin that separates clinically important from clinically negligible (acceptable) differences; p = 0.89, Mixed Models Analysis; Mean Difference (Net) = -0.09, 95% CI 2-sided [-1.35 to 1.17], Standard Deviation 1.26

5. Primary Outcome: Depression, as Assessed by Hamilton Depression Rating Scale(Ham-D)
Description: Ham-D indicates Hamilton Depression Rating Scale,range is 0 to 52. A score of 0 means the best outcome with no depression symptoms reported, and a score of 52 is the worse outcome with highest level of depression reported. A difference of 3 points on the Hamilton scale has been identified as clinically significant.
Time Frame: Measured at baseline; Weeks 4, 9, 14, and 18; and Months 3, 6, 9, and 12 of follow-up
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Telephone-administered CBT | Face-to-face CBT
Number analyzed (Participants) | 163 | 162
units on a scale
  Baseline | 22.83 (4.6) [22.34 to 23.33] | 22.83 (4.6) [22.34 to 23.33]
  Week04 | 18.07 [17.16 to 18.98] | 17.86 [16.96 to 18.77]
  Week09 | 15.62 [14.60 to 16.65] | 16.45 [15.40 to 17.51]
  Week14 | 14.94 [13.77 to 16.12] | 14.18 [12.97 to 15.39]
  Week18 | 13.58 [12.42 to 14.74] | 12.51 [11.22 to 13.81]
  3-month follow-up | 14.58 [13.45 to 15.71] | 12.33 [11.1 to 13.64]
  6-month follow-up | 15.06 [13.84 to 16.27] | 12.14 [10.84 to 13.45]
Statistical Analysis 1: Comparison: Telephone-administered CBT vs Face-to-face CBT; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p = 0.22, Mixed Models Analysis; Mean Difference (Net) = 1.07, 95% CI 2-sided [-0.63 to 2.76], Standard Deviation 1.695

ADVERSE EVENTS:
Arm/Group | Telephone-administered CBT | Face-to-face CBT
Serious Adverse Events (participants affected / at risk) | 0/163 | 0/162
Other Adverse Events (participants affected / at risk) | 0/163 | 0/162

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No